CLINICAL TRIAL: NCT02136680
Title: CASA: Care and Support Access Study for Implementation of a Palliative Approach With HIV Treatment
Brief Title: CASA: Care and Support Access in HIV Disease
Acronym: CASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); New York University (Other)
Responsible Party: Principal Investigator, Carla Alexander, Assistant Professor of Medicine, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HP-00058180
Record Dates: First submitted 2014-05-05; First posted 2014-05-13 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: HIV/AIDS
Keywords: HIV disease; palliative care; educational intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients at Intervention Site (Active Comparator): Staff receives CASA Education
  Interventions: Other: CASA Education
- Patients at CONTROL site (No Intervention): Staff does not receive CASA Education

INTERVENTIONS:
Other: CASA Education — Basic palliative care competencies for outpatient use.
  Arms: Patients at Intervention Site

SUMMARY:
This is an investigator-initiated study to measure the impact of an educational intervention on the basic palliative approach for a multidisciplinary staff team at an outpatient HIV clinic. The study aims to: 1) refine a curriculum for non-palliative care clinicians caring for persons living with HIV disease early in the disease trajectory; 2) assess the impact of the palliative approach educational intervention on outcomes for 2 target populations: a) patients (mental health, quality of life, health-related quality of life and secondarily, retention in care and viral suppression) and b) staff (burn-out and caregiving stress). It is hypothesized that training outpatient HIV staff in palliative care competencies will improve care provided that might, in turn, improve clinical outcomes for HIV patients receiving care at that clinic. Quantitative data will be augmented by qualitative interviews of selected staff and patients at both clinics in the final year of the study to appreciate response to the intervention.

DETAILED DESCRIPTION:
Evidence exists in African populations that palliative care delivered early in the HIV disease trajectory can improve symptom management and mental health. This study represents a proof of principle for HIV care delivery in the US using observed distillation of critical palliative elements.

Care and Support Access (CASA) is a complex multidisciplinary care strategy in which a palliative approach is integrated into the delivery of standard HIV care, using an iterative teaching method and on-site mentored training of site-based care teams. CASA will implement patient-centeredness into HIV treatment at the practice setting to improve patient-level outcomes for persons with HIV/AIDS known to have difficulty in engaging in care, initiating antiretroviral therapy (ART), and remaining in routine follow-up. This lack of retention puts them at high risk for experiencing health-related symptoms and poor quality of life (QOL).

The study design is quasi-experimental with longitudinal observation of the HIV positive young men who have sex with men (yMSM) population and staff who deliver their care at two HIV outpatient clinics. We use mixed methods (surveys and qualitative interviews) with the patients and staff at both clinics.

The Specific Aims are:

(1) To refine, deliver and determine the acceptability and applicability of an interdisciplinary professional education program for a site-based multidisciplinary health care team on the integration of basic palliative care domains fundamental to patient-centered care with standard HIV care.

2) To obtain insights regarding the CASA experience and to describe and measure the impact of early integration of a palliative approach upon yMSM relative to: a) improvement of mental health status, health-related quality of life and overall quality of life; b) increased retention in care and viral suppression.

3) To describe and measure the impact upon staff of the early integration of the palliative approach with regard to: a) reducing work-related stress; and b) burn-out.

The anticipated impact of the CASA study will be to improve clinical practice with regard to engagement and retention of difficult to engage and retain patient populations by introducing a basic palliative approach to care management.

ELIGIBILITY:
PATIENTS -

Inclusion Criteria:

* HIV positive
* men who have sex with men attending one of 2 study site clinics
* 18-35 years

Exclusion Criteria:

* acute illness requiring medical attention
* cognitive impairment

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The specific patient population being addressed in this study is HIV positive young men who have sex with men (yMSM). We are targeting HIV positive yMSM because they are at high risk for poor personal outcomes and are currently recognized as a significant barrier in efforts to prevent HIV infection in Baltimore, one of 20 US cities with high HIV prevalence.
Enrollment: 197 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla S Alexander, MD, Principal Investigator — University of Maryland School of Medicine-Institute of Human Virology; Victoria H Raveis, PhD, Principal Investigator — New York University, College of Dentistry - Psychosocial Research Unit on Health, Aging and the Community
Locations (1):
- University of Maryland Medical System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander CS, Pappas G, Amoroso A, Lee MC, Brown-Henley Y, Memiah P, O'Neill JF, Dix O, Redfield RR; Members of the AIDSRelief Consortium of PEPFAR. Implementation of HIV Palliative Care: Interprofessional Education to Improve Patient Outcomes in Resource-Constrained Settings, 2004-2012. J Pain Symptom Manage. 2015 Sep;50(3):350-61. doi: 10.1016/j.jpainsymman.2015.03.021. Epub 2015 Jul 16. PMID 26188088
- [Background] Alexander CS, Raveis VH, Karus DG, Lee MC, Tagle MC, Brotemarkle R, et al. Patient centered care for persons with HIV disease: Protocol review for CASA study (Care and Support Access) early in chronic disease management. Journal of Palliative Care & Medicine 7:300, 2017. doi: 10.4172/2165-7386.1000300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between July 2014 and June of 2016. Enrollment took place in 2 separate HIV outpatient clinics where most clinic attendees were known to be HIV positive.
Pre-assignment Details: Potential participants were identified initially by age and gender, recruited and, if eligible, retained as study participants. We solicited referrals of eligible patients from primary care providers or designated clinic staff, and reviewed appointment schedules at both sites. Initial contact was made by the participant's primary care provider.
Groups:
- Patients at Intervention Site: Staff receives CASA Education:
  The intervention is to deliver staff education and training for early integration of palliative skills with ongoing HIV management. Palliative skills for individuals who have little, or no, formal training in palliative care focus on care strategies to relieve suffering and promote quality of life for persons with any chronic illness regardless of the life expectancy. The educational intervention is based upon 8 years' experience in training clinicians how to care for HIV patients using a "Train the Trainer" method and quality improvement to integrate palliative skills with HIV care and treatment. The model used for this training is standard in chronic disease management and was used by the University of Maryland, Baltimore research team for 8 years in African settings. These skills can be applied to any chronic illness.
- Patients at CONTROL Site: Staff does not receive CASA Education:
  Patients at this site receive their usual care.
Period: Overall Study
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Started | 112 | 85
Interview 1 | 112 | 85
Interview 2 | 97 | 70
Interview 3 | 80 | 56
Completed | 80 | 56
Not Completed | 32 | 29
Not completed — No Longer Interested | 1 | 1
Not completed — No longer receiving care at clinic | 3 | 5
Not completed — Moved away | 5 | 4
Not completed — Unable to schedule | 17 | 16
Not completed — Study ended before interview due | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Patients at Intervention Site: Staff receives CASA Education: Basic palliative competencies for outpatient use.
- Total: Total of all reporting groups
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site | Total
Number analyzed (Participants) | 112 | 85 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (4.2) | 30 (3.5) | 29 (3.9)
Age, Customized [Count of Participants; unit: Participants]
  18 - 25 | 29 | 11 | 40
  26 - 30 | 44 | 39 | 83
  31 - 35 | 39 | 35 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 112 | 85 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Hispanic | 93 | 61 | 154
  Hispanic | 11 | 7 | 18
  White, non-Hispanic | 2 | 9 | 11
  Other, non-Hispanic | 0 | 4 | 4
  Multiracial, non-Hispanic | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 85 | 197
HIV Risk Group [Count of Participants; unit: Participants] — Perceived mode of HIV transmission Population: There was insufficient information to categorize 2 participants.
  Participants
    number analyzed (Participants) | 110 | 85 | 195
    Sex | 89 | 63 | 152
    Sex (Female Only) | 3 | 0 | 3
    IV Drug Usage | 2 | 1 | 3
    Transfusion | 1 | 0 | 1
    Sex and IV Drug Usage | 2 | 6 | 8
    Sex, IV Drug Usage and Transfusion | 9 | 7 | 16
    Other | 1 | 1 | 2
    Don't know | 3 | 7 | 10
IV Drug Usage Risk Factor [Count of Participants; unit: Participants] — Participant risk factor for IV drug usage. Population: There was insufficient information to categorize 2 participants.
  Participants
    number analyzed (Participants) | 110 | 85 | 195
    No | 97 | 71 | 168
    Yes | 13 | 14 | 27
HIV Treatment Regimen [Count of Participants; unit: Participants] — Number of pills taken.
  Participants
    No Treatment | 1 | 1 | 2
    1 Pill/Day | 91 | 53 | 144
    2 or More Pills/Day | 19 | 28 | 47
    No Medical Info | 1 | 3 | 4
Viral Load Suppressed [Count of Participants; unit: Participants] — Participant is HIV viral load suppressed.
  Participants
    Unknown | 16 | 4 | 20
    No | 39 | 31 | 70
    Yes | 57 | 50 | 107
Adherence [Count of Participants; unit: Participants] — Self-reported adherence over the past month by an item from the Adult Aids Clinical Trials Group (AACTG) questionnaire.
  Participants
    Not adherent | 53 | 39 | 92
    Adherent | 59 | 45 | 104
    Missing Info | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mental Health: Rosenberg Self-Esteem Scale
Description: Rosenberg Self-Esteem Scale: The Rosenberg Self-Esteem Scale (RSES) is a 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is well validated and has been used in a wide variety of populations, including persons living with HIV/AIDS. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree. Scores for individual items varied in range from 1 to 4, with higher scores indicative of greater self-esteem. Summary score is reflective of the mean score across all items.
Time Frame: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Population: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Measure: Mean (Standard Deviation); unit: [Units on a scale]
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Number analyzed (Participants) | 112 | 85
[Units on a scale]
  Baseline | 3.2 (0.6) | 3.2 (0.6)
  FU1: number analyzed (Participants) | 97 | 70
  FU1 | 3.2 (0.5) | 3.1 (0.6)
  FU2: number analyzed (Participants) | 80 | 56
  FU2 | 3.1 (0.6) | 3.0 (0.6)
Statistical Analysis 1: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Self-Esteem from Baseline to First Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.400, Regression, Linear; Regression Coefficient = 0.046
Statistical Analysis 2: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Self-Esteem from Baseline to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.022, Regression, Linear; Regression Coefficient = 0.119
Statistical Analysis 3: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Self-Esteem from First Follow-up to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.347, Regression, Linear; Regression Coefficient = -0.003

2. Primary Outcome: Quality of Life: McGill Quality of Life Scale
Description: The McGill Quality of Life Questionnaire (MQOL) is a measure of quality of life for persons with advanced/serious illness. The MQOL consists of 16-items plus a global quality of life item, each with a 2-day time frame and has demonstrated validity and other measurement properties for use with palliative care populations. There are four subscales (psychological symptoms, existential well-being, support, and physical symptoms) and a summary quality of life score that weights these domains equally. Items are scored zero (worst) to 10 (excellent).
Time Frame: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Population: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Measure: Mean (Standard Deviation); unit: [Units on a scale]
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Number analyzed (Participants) | 112 | 85
[Units on a scale]
  Baseline: Global QOL Item | 6.9 (2.4) | 6.7 (2.6)
  Baseline: Summary QOL Score | 7.0 (2.1) | 6.9 (2.1)
  FU1: Global QOL Item: number analyzed (Participants) | 97 | 85
  FU1: Global QOL Item | 7.3 (2.3) | 7.1 (2.5)
  FU1: Summary QOL Score: number analyzed (Participants) | 97 | 70
  FU1: Summary QOL Score | 7.0 (2.2) | 6.9 (2.3)
  FU2: Global QOL Item: number analyzed (Participants) | 80 | 85
  FU2: Global QOL Item | 7.2 (2.5) | 6.4 (2.8)
  FU2: Summary QOL Score: number analyzed (Participants) | 80 | 56
  FU2: Summary QOL Score | 7.1 (2.3) | 6.2 (2.2)
Statistical Analysis 1: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Global QOL from Baseline to First Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.959, Regression, Linear; Regression Coefficient = -0.003
Statistical Analysis 2: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Global QOL from Baseline to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.021, Regression, Linear; Regression Coefficient = 0.143
Statistical Analysis 3: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Global QOL from First Follow-up to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.454, Regression, Linear; Regression Coefficient = 0.048
Statistical Analysis 4: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Summary QOL from Baseline to First Follow-up; Test type: Superiority; p = 0.774, Regression, Linear; Regression Coefficient = -0.015
Statistical Analysis 5: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Summary QOL from Baseline to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.018, Regression, Linear; Regression Coefficient = 0.137
Statistical Analysis 6: Comparison: Patients at Intervention Site; Change in Summary QOL from First Follow-up to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.362, Regression, Linear; Regression Coefficient = 0.051

3. Primary Outcome: Health-Related Quality of Life in Palliative Care: Palliative Outcome Scale
Description: The Palliative Outcome Scale (POS) is a 10-item multidimensional well-being tool well validated for use in palliative care settings that measures the 3-day period prevalence and intensity of pain, other physical symptoms, patient anxiety, family/friends anxiety, information sufficiency, sharing feelings with family/friends, feeling life is worthwhile, self-worth, wasted time, and personal affairs, i.e. the physical/social/spiritual/psychological problems in line with the World Health Organization (WHO) definition of palliative care. Eight of the 10 items use a five-point Likert-like scale, and the remaining two items use a three-point scale. Scores for respondents' ratings on all items can range from 0 (indicating no problem) to 4 (indicating a very severe or overwhelming problem). The overall profile score is the sum of the scores from each of the 10 questions and can therefore range from zero to 40. Higher scores are indicative of greater problems.
Time Frame: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Population: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Measure: Mean (Standard Deviation); unit: [Units on a scale]
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Number analyzed (Participants) | 112 | 85
[Units on a scale]
  Baseline | 8.9 (7.0) | 8.4 (6.6)
  FU1: number analyzed (Participants) | 97 | 69
  FU1 | 8.4 (6.4) | 9.5 (7.0)
  FU2: number analyzed (Participants) | 80 | 55
  FU2 | 8.5 (7.1) | 8.5 (6.5)
Statistical Analysis 1: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Palliative Outcomes from Baseline to First Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.213, Regression, Linear; Regression Coefficient = -0.072
Statistical Analysis 2: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Change in Palliative Outcomes from Baseline to Second Follow-up: Intervention Group vs. Control Group; Test type: Superiority; p = 0.561, Regression, Linear; Regression Coefficient = 0.037
Statistical Analysis 3: Comparison: Patients at Intervention Site vs Patients at CONTROL Site; Test type: Superiority — Change in Palliative Outcomes from First Follow-up to Second Follow-up: Intervention Group vs. Control Group; p = 0.008, Regression, Linear; Regression Coefficient = 0.165

4. Secondary Outcome: Viral Load Suppressed
Description: Patient is HIV viral load suppressed, as abstracted from patient electronic medical records.
Time Frame: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Population: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1. There were 11 cases for which viral load information was missing from the patient medical records.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Number analyzed (Participants) | 102 | 84
Participants
  Baseline: Not Virally Suppressed | 43 | 32
  Baseline: Viral Load Suppressed | 59 | 52
  FU1: number analyzed (Participants) | 73 | 64
  FU1: Not Virally Suppressed | 25 | 20
  FU1: Viral Load Suppressed | 48 | 44
  FU2: number analyzed (Participants) | 68 | 55
  FU2: Not Virally Suppressed | 18 | 19
  FU2: Viral Load Suppressed | 50 | 36

5. Secondary Outcome: Adherence
Description: Self-reported adherence over the past month by an item from the Adult Aids Clinical Trials Group (AACTG) questionnaire.
Time Frame: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1
Population: Baseline, 1st Follow-up [FU1]: 4-5 mos post-initiation of baseline/intervention, 2nd Follow-up [FU2]: 4-5 mos post FU1. There was 1 case for which adherence data was missing for the patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
Number analyzed (Participants) | 112 | 84
Participants
  Baseline: Not Adherent | 53 | 39
  Baseline: Adherent | 59 | 45
  FU1: number analyzed (Participants) | 97 | 70
  FU1: Not Adherent | 42 | 41
  FU1: Adherent | 55 | 29
  FU2: number analyzed (Participants) | 80 | 55
  FU2: Not Adherent | 34 | 33
  FU2: Adherent | 46 | 22

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Groups:
- Patients at Intervention Site: Staff receives CASA Education
  CASA Education: Basic palliative competencies for outpatient use.
Arm/Group | Patients at Intervention Site | Patients at CONTROL Site
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/85
Other Adverse Events (participants affected / at risk) | 0/112 | 0/85

LIMITATIONS AND CAVEATS:
Due to the duration of the study, while it was feasible to obtain short-term follow-up of participants, it was not possible because of an extension of the recruitment period to obtain long-term follow-up data on the complete panel sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form: Patient Informed Consent Form (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT02136680/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02136680/Prot_SAP_001.pdf
  • Informed Consent Form: Staff Informed Consent Form (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02136680/ICF_002.pdf